CLINICAL TRIAL: NCT01863537
Title: Using Multimedia Technologies to Disseminate an HIV Prevention Program for Couples
Brief Title: Using Multimedia Technologies to Disseminate an HIV Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Susan Witte, Associatge Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AAAC5642; R01MH080659 (NIH)
Record Dates: First submitted 2013-05-20; First posted 2013-05-29 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Multimedia Connect and the Multimedia facilitator training curriculum with a 4-day, face-to-face structured orientation and training for implementation, and planned, investigative team initiated telephone consultations with CBO staff to provide technical assistance at 2 and 4 months following the training workshop;
  Interventions: Behavioral: Multimedia Connect
- Traditional Connect (Active Comparator): The original, manualized version of Connect (CDC DEBI)and manualized facilitator training curriculum with a 4-day, face-to-face structured orientation and training for implementation, and planned, investigative team initiated telephone consultation with CBO staff to provide technical assistance at 2 and 4 months following the training workshop.
  Interventions: Behavioral: Traditional Connect

INTERVENTIONS:
Behavioral: Multimedia Connect
  Arms: Intervention
Behavioral: Traditional Connect
  Arms: Traditional Connect

SUMMARY:
This RCT will randomly assign 40 of the CBOs to receive the Multimedia intervention and training package (Multimedia)and the other 40 to receive the original, manualized Connect intervention and training package (Traditional). The technology transfer process involves all agencies receiving four days of training and two planned technical assistance conference calls, by study investigative staff, in the first four months following training. Telephone assessments completed by up to 6 staff at each agency will measure primary outcomes, mediating, moderating and process measure variables at baseline, 6, 12 and 18 months post-technology transfer. The primary outcome of the study is adoptions of the Connect intervention. The unit of analysis is the CBO.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, CBOs must have reported that they

* had 501c3 status;
* provided at least a minimum level of direct contact HIV prevention services to clientele; and
* that their target population for services included heterosexual men and women.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2007-05; Primary Completion 2011-09 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The mean number of Connect sessions per client/couple implemented by participating staff (at each agency) in the prior 6 months | 18 months

SECONDARY OUTCOMES:
To test whether key variables mediate adoption outcomes (e.g. staff attitudes and opinions towards programming and technology). | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan S. Witte, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Social Intervention Group, New York, New York, United States

REFERENCES:
- [Derived] Witte SS, Wu E, El-Bassel N, Hunt T, Gilbert L, Medina KP, Chang M, Kelsey R, Rowe J, Remien R. Implementation of a couple-based HIV prevention program: a cluster randomized trial comparing manual versus Web-based approaches. Implement Sci. 2014 Sep 11;9:116. doi: 10.1186/s13012-014-0116-x. PMID 25208569